CLINICAL TRIAL: NCT01064102
Title: Experimental Evaluation of Relative Bioavailabilities of Two Formulations of Cetirizine Hydrochloride Tablets 10 mg in Healthy Adult Human Male Subjects Under Fasting Conditions.
Brief Title: Cetirizine Hydrochloride Tablets, 10 mg Bioequivalence Study of Dr.Reddy's Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Senior Manager - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 007-06
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
MeSH Terms: interventions — Cetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetirizine (Experimental): Cetirizine Hydrochloride Tablets 10 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Cetirizine Hydrochloride
- Zyrtec (Active Comparator): Zyrtec Tablets 10 mg of Pfizer Labs
  Interventions: Drug: Cetirizine Hydrochloride

INTERVENTIONS:
Drug: Cetirizine Hydrochloride — Cetirizine Hydrochloride Tablets 10 mg
  Other Names: Zyrtec Tablets 10 mg

SUMMARY:
A Two Way, Open Label, Single Dose, Cross Over, Experimental Evaluation of Relative Bioavailabilities of Two Formulations of Cetirizine Hydrochloride Tablets 10 mg of Dr. Reddys laboratories with Zyrtec 10 mg of Pfizer labs in Healthy Adult Human Male Subjects Under Fasting Conditions.

DETAILED DESCRIPTION:
Open Label, Balanced, Randomized, Two-Treatment, Two-Period, Two-Sequence, Single Dose, Cross Over, and Comparative Oral Bioavailability study in healthy, adult, human, male subjects under Fasting Conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between 18 and 45 years of age (both inclusive) living in and around Ahmedabad city of western part of India.
2. Having a Body Mass Index (BMI) between 18.5 and 24.9 {both inclusive), calculated as weight in kg/height in m2
3. Not having any significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, ECG and X-ray recordings.
4. Able to comply with the study procedures, in the opinion of the investigator.
5. Able to give written consent for participation in the trial.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to cetirizine or any other related drugs.
2. Any disease or condition which might compromise the hemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
3. Use of any medicine within 14 days prior to start of the study. In any such case subject selection will be at the discretion of the Principal investigator / Medical expert
4. Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
5. A recent history of alcoholism (<2 years) or of moderate (180 mL/day) alcohol use, or consumption of alcohol within 48 hr prior to receiving IP.
6. Smokers, who smoke more than 10 cigarettes / day or inability to abstain from smoking during the study.
7. The presence of clinically significant abnormal laboratory values during screening.
8. Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
9. History of psychiatric disorders.
10. A history of difficulty in donating blood.
11. Donation of blood (1 unit or 350 mL) within 90 days prior to receiving the first dose of IP.

    Note: In case, the blood loss was ≤200 mL; subject can be dosed 60 days after the blood donation.
12. A positive hepatitis screen including hepatitis B surface antigen, Anti- HCV and Anti HAV antibodies.
13. A positive test result for HIV antibody and/or syphilis.
14. The receipt of an investigational drug or product, or participation in a drug research study within a period of 90 days prior to the first dose of IP (Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study).

    Note: If subject had participated in a study in which blood loss was ≤200 mL, subject can be dosed after completion of 60 days after the last sample of the previous study.
15. An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the IP and throughout the subjects participation in the study. In any such case subject selection will be at the discretion of the Principal lnvestigator/Medical expert.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Bio-equivalence study of Dr Reddys Laboratories Cetirizine Hydrochloride Tablets 10 mg | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Charu Gautam, MD, Principal Investigator — Lambda Therapeutic Research Ltd, Ahmedabad - 380 054, Gujarat, INDIA